CLINICAL TRIAL: NCT00256126
Title: A Phase IV Open-label Study of Predictive Markers in Growth Hormone Deficient and Turner Syndrome Pre-pubertal Children Treated With SAIZEN®
Brief Title: Predictive Markers in Growth Hormone Deficiency (GHD) and Turner Syndrome (TS) Children Treated With SAIZEN®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24531
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: Growth Hormone Deficiency; Turner Syndrome
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome | interventions — Human Growth Hormone

ARMS (2):
- Turner Syndrome (TS) (Experimental)
  Interventions: Drug: Saizen
- Growth Hormone Deficiency (GHD) (Experimental)
  Interventions: Drug: Saizen

INTERVENTIONS:
Drug: Saizen — Subjects with TS will receive SAIZEN® as subcutaneous injection at a dose of 0.050 milligram per kilogram (mg/kg) of body weight per day (within the recommended dosage 0.045-0.050 mg/kg body weight) for a period of 1 month
  Arms: Turner Syndrome (TS)
Drug: Saizen — Subjects with GHD will receive SAIZEN® as subcutaneous injection at a dose of 0.035 mg/kg of body weight per day (within the recommended dosage 0.025-0.035 mg/kg body weight) for a period of 1 month.
  Arms: Growth Hormone Deficiency (GHD)

SUMMARY:
The study aims at identifying the predictive markers after one month of Saizen therapy in Growth Hormone Deficiency (GHD) and Turner Syndrome children.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses and candidacy for SAIZEN® therapy:

A) GHD: documented pre-established diagnosis of GHD with a growth hormone (GH) peak response of <10 microgram per liter (mcg/L) with 2 GH stimulation tests, without priming with oestradiol.

B) Turner syndrome: documented pre-established diagnosis by karyotype.

* Prepubertal status according to Tanner Pre-established history of normal thyroid function or adequate substitution for at least 3 months.
* Weight for stature within the population specific normal range (>5th and <95th percentiles) for gender Willingness and ability to comply with the protocol for the duration of the study.
* Parent's or guardian's written informed consent, given before any study related procedure that is not part of the subject's normal medical care, with the understanding that the subject or parent/guardian may withdraw consent at any time without prejudice to future medical care. If the child is old enough to read and write, a separate assent form will be given.

Exclusion Criteria:

* Acquired GHD due to central nervous system tumour, trauma, infection, infiltration (documented by imaging), and history of irradiation or cranial surgery
* Previous treatment with GH, growth hormone-releasing hormone (GHRH), anabolic steroids or any treatment affecting growth.
* Previous treatment with corticosteroids, except in case of topical or inhaled corticosteroid administration for atopic disease. Corticosteroids for hormonal substitution are also allowed if the condition and the treatment regimen have been stable for at least 3 months.
* Severe associated pathology affecting growth such as malnutrition, malabsorption, or bone dysplasia.
* Chronic severe kidney disease.
* Chronic severe liver disease.
* Chronic infectious disease.
* Acute or severe illness during the previous 6 months.
* Significant concomitant illness that would interfere with participation or assessment in this study.
* Active malignancy (except non-melanomatous skin malignancies that have undergone surgical excision and/or biopsy, diagnosis and treatment to resolution)
* History or active Idiopathic intra-cranial hypertension (benign intracranial hypertension or pseudo-tumor cerebri).
* Diabetes Mellitus type I & II.
* Any autoimmune disease.
* Previous screening failure in this study.
* Use of an investigational drug or participation in another clinical study within the last three months.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2005-05-31 (Actual); Primary Completion 2007-09-30 (Actual); Study Completion 2007-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (13):
- Local Medical Information Office, Buenos Aires, Argentina
- Local Medical Information Office, Sydney, Australia
- Local Medical Information Office, Vienna, Austria
- Local Medical Information Office, Mississauga, Canada
- Local Medical InformationOffice, Paris, France
- Local Medical Information Office, Munich, Germany
- Local Medical Information Office, Rome, Italy
- Local Medical Information Office, Oslo, Norway
- Local Medical Information Office, Russia, Russia
- Local Medical Information Office, Singapore, Singapore
- Local Medical Information Office, Madrid, Spain
- Local Medical Information Office, Stockholm, Sweden
- Local Medical Information Office, Feltham, United Kingdom

REFERENCES:
- [Result] Stevens A, Clayton P, Tato L, Yoo HW, Rodriguez-Arnao MD, Skorodok J, Ambler GR, Zignani M, Zieschang J, Della Corte G, Destenaves B, Champigneulle A, Raelson J, Chatelain P. Pharmacogenomics of insulin-like growth factor-I generation during GH treatment in children with GH deficiency or Turner syndrome. Pharmacogenomics J. 2014 Feb;14(1):54-62. doi: 10.1038/tpj.2013.14. Epub 2013 Apr 9. PMID 23567489
- [Derived] Stevens A, Murray P, De Leonibus C, Garner T, Koledova E, Ambler G, Kapelari K, Binder G, Maghnie M, Zucchini S, Bashnina E, Skorodok J, Yeste D, Belgorosky A, Siguero JL, Coutant R, Vangsoy-Hansen E, Hagenas L, Dahlgren J, Deal C, Chatelain P, Clayton P. Gene expression signatures predict response to therapy with growth hormone. Pharmacogenomics J. 2021 Oct;21(5):594-607. doi: 10.1038/s41397-021-00237-5. Epub 2021 May 27. PMID 34045667
- [Derived] Murray PG, Stevens A, De Leonibus C, Koledova E, Chatelain P, Clayton PE. Transcriptomics and machine learning predict diagnosis and severity of growth hormone deficiency. JCI Insight. 2018 Apr 5;3(7):e93247. doi: 10.1172/jci.insight.93247. eCollection 2018 Apr 5. PMID 29618660
- [Derived] Valsesia A, Chatelain P, Stevens A, Peterkova VA, Belgorosky A, Maghnie M, Antoniazzi F, Koledova E, Wojcik J, Farmer P, Destenaves B, Clayton P; PREDICT Investigator group. GH deficiency status combined with GH receptor polymorphism affects response to GH in children. Eur J Endocrinol. 2015 Dec;173(6):777-89. doi: 10.1530/EJE-15-0474. Epub 2015 Sep 4. PMID 26340968
- See also: Full FDA approved prescribing information can be found here — http://www.saizenus.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First informed consent date: May 2005. Clinical data cutoff date: Oct 2007, Study completion date: Sep 2007.
Pre-assignment Details: A total of 319 subjects were screened for this trial. Only 1 subject withdrew from the study prior to receiving the treatment due to personal reasons. Overall, 318 subjects were enrolled into the study.
Groups:
- Turner Syndrome (TS): Subjects with TS were administered with SAIZEN® as subcutaneous injection at a dose of 0.050 milligram per kilogram (mg/kg) of body weight per day (within the recommended dosage 0.045-0.050 mg/kg body weight) for a period of 1 month.
- Growth Hormone Deficiency (GHD): Subjects with GHD were administered with SAIZEN® as subcutaneous injection at a dose of 0.035 mg/kg of body weight per day (within the recommended dosage 0.025-0.035 mg/kg body weight) for a period of 1 month.
Period: Overall Study
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Started | 149 | 169
Completed | 147 | 167
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD) | Total
Number analyzed (Participants) | 149 | 169 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.08) | 8.94 (3.17) | 9.11 (3.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 63 | 212
  Male | 0 | 106 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Like Growth Factor-1 Standard Deviation Score (IGF-1 SDS) at Month 1
Description: IGF-1 SDS was calculated using the Elmlinger reference method. Change in within subject IGF-1 levels (standard deviation scores) at Month 1 from Baseline was assessed. Descriptive statistics were determined for the Baseline and Month 1 assessments, and also for the level of change between these two assessments. If either the Baseline or Month 1 IGF-1 level was missing, then the within-subject change in IGF-1 was assumed to be missing.
Time Frame: Baseline, Month 1
Population: The Intention to Treat (ITT) population included all subjects who received at least 1 dose of study medication. Here "Overall Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Standard deviation score (SDS)
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 143 | 162
Standard deviation score (SDS) | 1.7692 (1.1889) | 1.4007 (0.9811)
Statistical Analysis 1: Comparison: Turner Syndrome (TS) vs Growth Hormone Deficiency (GHD); Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor Binding Protein - 3 (IGFBP-3) Level at Month 1
Time Frame: Baseline, Month 1
Population: The ITT population included all subjects who received at least 1 dose of study medication. Here "Overall Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 143 | 162
milligram per liter (mg/L) | 0.86 (0.96) | 0.69 (0.81)

3. Secondary Outcome: Change From Baseline in Fasting Glucose Levels at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 122 | 142
millimoles per liter (mmol/L) | 0.22 (0.8) | 0.13 (0.65)

4. Secondary Outcome: Change From Baseline in Fasting Insulin Levels at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 142 | 160
picomole per liter (pmol/L) | 47.7 (177.2) | 26.9 (79.8)

5. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) at Month 1
Description: HOMA-IR is used to assess insulin resistance and calculated by an empirical mathematical formula based on fasting plasma glucose and fasting plasma insulin levels. HOMA-IR = fasting plasma insulin (picomole/liter [pmol/L]) * fasting plasma glucose (millimole/liter [mmol/L]) divided by 22.5.
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomole per liter *millimole per liter
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 120 | 136
picomole per liter *millimole per liter | 2.132 (10.296) | 1.061 (3.885)

6. Secondary Outcome: Change From Baseline in Bone Alkaline Phosphatase Levels at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Number analyzed (Participants) | 144 | 162
Units per liter (U/L) | 21.13 (80.68) | 14.78 (25.23)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from first dose until at least 4 weeks following the last SAIZEN® administration or the post-treatment visit, whichever represented the longer period (up to a maximum of 2 months).
Arm/Group | Turner Syndrome (TS) | Growth Hormone Deficiency (GHD)
Serious Adverse Events (participants affected / at risk) | 0/149 | 1/169
Other Adverse Events (participants affected / at risk) | 36/149 | 51/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turner Syndrome (TS) (N=149) | Growth Hormone Deficiency (GHD) (N=169)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turner Syndrome (TS) (N=149) | Growth Hormone Deficiency (GHD) (N=169)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 9 (9)
Injection site haemorrhage (General disorders) | 1 (1) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site anaesthesia (General disorders) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 12 (18)
Dizziness (Nervous system disorders) | 2 (3) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Precocious puberty (Endocrine disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (2) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial were short duration of the study treatment, and relatively small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other